CLINICAL TRIAL: NCT03661203
Title: The Issue of Late Recourse to HIV Testing. A Study of the Psychosocial Factors at Play Within Men Who Have Sex With Men in France.
Brief Title: Investigation of the Psychosocial Factors Responsible for the Late Recourse to HIV Testing Within MSM
Acronym: ReTarD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: University of Lyon (Other)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Other Study IDs: ANRS ReTarD VIH; 2018-A00825-50 (Other: French FDA Registration Number (ANSM))
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-01

CONDITIONS: AIDS; HIV Seropositivity
Keywords: MSM population; Hindrances HIV screening; Late recourse HIV test; Healt social psychology
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Seropositivity | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Qualitative cohort: The cohort consists of MSM with late HIV diagnosis. The person from this cohort will participate to round table called also focus group or individual interview.
  Interventions: Behavioral: Focus group; Behavioral: Individual interview; Behavioral: self questionnaire
- Quantitative cohort: MSM community will be invited to participate to an online self questionnaire established from the information gathered from the previous cohort.
  Interventions: Behavioral: online self questionnaire

INTERVENTIONS:
Behavioral: Focus group — Focus group for qualitative group only
  Groups: Qualitative cohort
Behavioral: Individual interview — Individual interview for qualitative group only
  Groups: Qualitative cohort
Behavioral: online self questionnaire — online self questionnaire
  Groups: Quantitative cohort
Behavioral: self questionnaire — online self questionnaire following focus group or individual interview For qualitative group only
  Groups: Qualitative cohort

SUMMARY:
The present study will try to investigate and analyze the psycho-social hindrances and levers concerning the recourse to late HIV testing among the MSM population.

This study is divided in two parts. The first one will consist of individual and groups interviews. Then, depending on the items that will rise from the first part of the study, groups interview will take place based on theses items. Finally, a questionnaire build from the collected information will be sent to MSM community in order to obtain quantitative results.

DETAILED DESCRIPTION:
The late recourse to HIV testing, among the population in general way and among MSM population in a more specific way, participates in the dissemination of the HIV epidemic. Actually, there is no cure for HIV infection, but treatments that reduce viral charge to undetectable level exists. When diagnosed and treated earlier, seropositive people will be less communicating the virus because of the reduction of their viral charge.

This study aims to uncover the reasons behind the late recourse to HIV testing in MSM population facing a high risk of contamination.

The study hypothesis, is that late recourse to HIV testing is probably related to social and economics factors like age, social standing, accessibility to the diagnosis or even to a traditional beliefs or a fear of stigma etc. To shed the light on these factors, the main objectives of the investigator will try to investigate and analyze the psycho-social hindrances and levers through a quantitative and qualitative approach. This plurality of approaches is a part of a methodological triangulation method described by Kalampalikis & Apostolidis, 2016.

People among MSM community having had a late or very late HIV test (as defined by biological parameters :CD4≤200/mm3 or having been diagnosed with AIDS), will be recruited in this study. During the first phase of the study, the eligible population will participate to individual or group interview . This qualitative part of the project will allow the set up of a questionnaire that will be diffused widely to the MSM community to have quantitative results.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive
* Self-reported homo-or bisexual contamination mode
* TCD4 + / mm3 200 200 lymphocyte count or Have an AIDS classifying event
* Diagnosis of HIV positive for at least two months and for a maximum of 24 months

Exclusion Criteria:

* Primary infection

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-determination
Study Population: MSM: men who have sex with men.
Sampling Method: Non-Probability Sample
Enrollment: 1190 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Socio-representational elements associated with the very late use of the HIV test | 3 years
  Imbrication of representations and tests related to HIV

SECONDARY OUTCOMES:
Means of risk management | 3 years
  Use of screening in the management of the risk of seroconversion
Representation and Knowledge of prevention methods | 3 years
  To understand the links between the different uses or non-uses of the biomedical prevention methods TasP (Treatment as Prevention), PrEP (Pre-Exposure Prohylaxis) and the methods of recourse to the screening test.
Sense of community belonging | 3 years
  Understand the interaction links between community belonging and the use of the screening test.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Préau, PR, Principal Investigator — Université Lumière Lyon 2
Locations (4):
- France (4):
  - Le 190, Paris
  - Hopital Saint-Antoine, Paris
  - Hôpital Pitié-Salpêtrière, Paris
  - Hôpital Bichat Claude-Bernard, Paris

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mabire-Yon R, Di Ciaccio M, Picard H, Palich R, Supervie V, Preau M. Psychosocial factors involved in the very infrequent use of HIV testing among French MSM: a cross-sectional study. Int J STD AIDS. 2023 Aug;34(9):603-607. doi: 10.1177/09564624231155762. Epub 2023 Feb 16. PMID 36798044